CLINICAL TRIAL: NCT00677807
Title: A 26-week Extension to a 26-week Treatment, Multicenter, Randomized, Double-blind, Placebo-controlled, Adaptive, Seamless, Parallel-group Study to Assess Safety, Tolerability and Efficacy of Two Doses of Indacaterol (150 and 300 µg o.d.) in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Safety, Tolerability and Efficacy of Indacaterol in Patients With Moderate-to-severe Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CQAB149B2335SE; 2008-000663-42 (EudraCT Number)
Record Dates: First submitted 2008-05-13; First posted 2008-05-15 (Estimated); Results first posted 2011-08-18 (Estimated); Last update posted 2011-08-22 (Estimated); Status verified 2011-08

CONDITIONS: COPD
Keywords: COPD; adults; β2-agonist; indacaterol
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — indacaterol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Indacaterol 150 µg (Experimental): Indacaterol 150 µg once-daily (o.d.) via single-dose dry-powder inhaler (SDDPI).
  The short acting (beta) β2-agonist (SABA) salbutamol/albuterol was available for rescue use throughout the study.
  Interventions: Drug: Indacaterol
- Indacaterol 300 µg (Experimental): Indacaterol 300 µg once-daily (o.d.) via single-dose dry-powder inhaler (SDDPI).
  The short acting (beta) β2-agonist (SABA) salbutamol/albuterol was available for rescue use throughout the study.
  Interventions: Drug: Indacaterol
- Placebo (Placebo Comparator): Placebo once-daily (o.d.) via SDDPI.
  The short acting (beta) β2-agonist (SABA) salbutamol/albuterol was available for rescue use throughout the study.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Indacaterol — Indacaterol once-daily (o.d.) via single-dose dry-powder inhaler (SDDPI)
  Arms: Indacaterol 150 µg; Indacaterol 300 µg
Drug: Placebo — Placebo once-daily (o.d.) via single-dose dry-powder inhaler (SDDPI)
  Arms: Placebo

SUMMARY:
This study evaluated the 1 year safety, tolerability and efficacy of indacaterol against placebo in the treatment of Chronic Obstructive Pulmonary Disease (COPD) patients

ELIGIBILITY:
Inclusion Criteria:

* Patients eligible to participate in the study extension, by definition, will have met the inclusion and exclusion criteria for the core 26 weeks and not met the withdrawal criteria for the core study B2335S at Visit 14 (the last visit of the core study B2335S and the first visit of the extension study B2335SE).
* In addition the following inclusion/exclusion criteria specified below must be met.

  1. Patients must complete Stage 2 of the core study B2335S (NCT00463567).
  2. Written informed consent to participate in the extension must be obtained.
  3. Patients must be able to comply with all study requirements.

Exclusion Criteria:

* Patients who were randomized to open-label tiotropium in Study B2335S.
* Patients who participated in Stage 1 of the core study (B2335S).
* Patients discontinued irrespective of the reason from Stage 2 of the core study.
* Patients who fail to comply with the core protocol requirements and procedures.
* Concomitant medical conditions that may interfere with interpretation of study results as defined in the core study protocol.
* Patients who in the Investigator's opinion should not participate in the extension study.

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 415 (Actual)
Dates: Start 2008-05; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (183):
- United States (86):
  - Novartis Investigative Site, Homewood, Alabama
  - Novartis Investigative Site, Jasper, Alabama
  - Novartis Investigative Site, Phoenix, Arizona
  - Novartis Investigative Site, Tucson, Arizona
  - Novartis Investigative Site, Pine Bluff, Arkansas
  - Novartis Investigative Site, Encinitas, California
  - Novartis Investigative SIte, Fullerton, California
  - Novartis Investigative Site, Orange, California
  - Novartis Investigative Site, Riverside, California
  - Novartis Investigative Site, Spring Valley, California
  - Novartis Investigative site, Fort Collins, Colorado
  - Novartis Investigative site, Golden, Colorado
  - Novartis Investigative Site, Wheat Ridge, Colorado
  - Novartis Investigative Site, Clearwater, Florida
  - Novartis Investigative Site, Largo, Florida
  - Novartis Investigative Site, Pensacola, Florida
  - Novartis Investigative Site, Rockledge, Florida
  - Novartis Investigative Site, South Miami, Florida
  - Novartis Investigative Site, Tamarac, Florida
  - Novartis Investigative Site, Tampa, Florida
  - Novartis Investigative Site, Atlanta, Georgia
  - Novartis Investigative Site, Marietta, Georgia
  - Novartis Investigative Site, Normal, Illinois
  - Novartis Investigative Site, O'Fallon, Illinois
  - Novartis Investigative Site, River Forest, Illinois
  - Novartis Investigative Site, Indianapolis, Indiana
  - Novartis Investigative Site, Iowa City, Iowa
  - Novartis Investigative Site, Topeka, Kansas
  - Novartis Investigative Site, Crescent Springs, Kentucky
  - Novartis Investigative Site, Lexington, Kentucky
  - Novartis Investigative Site, Lafayette, Louisiana
  - Novartis Investigative Site, Metaire, Louisiana
  - Novartis Investigative site, New Orleans, Louisiana
  - Novartis Investigative Site, Biddeford, Maine
  - Novartis Investgative Site, Clarkston, Michigan
  - Novartis Investigative Site, Flint, Michigan
  - Novartis Investigative Site, Livonia, Michigan
  - Novartis Investigative site, Troy, Michigan
  - Novartis Investigative Site, Minneapolis, Minnesota
  - Novartis Investigative Site, Rochester, Minnesota
  - Novartis Investigative Site, Chesterfield, Missouri
  - Novartis Investigative Site, Columbia, Missouri
  - Novartis Investigative Site, Kansas City, Missouri
  - Novartis Investigative Site, St Louis, Missouri
  - Novartis Investigative Site, Billings, Montana
  - Novartis Investigative Site, Kalispell, Montana
  - Novartis Investigative Site, Lincoln, Nebraska
  - Novartis Investigative Site, Omaha, Nebraska
  - Novartis Investigative Site, Papillion, Nebraska
  - Novartis Investigative site, Henderson, Nevada
  - Novartis Investigative site, Summit, New Jersey
  - Novartis Investigative Site, Elmira, New York
  - Novartis Investigative site, New York, New York
  - Novartis Investigative Site, Rochester, New York
  - Novartis Investigative Site, Charlotte, North Carolina
  - Novartis Investigative Site, Shelby, North Carolina
  - Novartis Investigative Site, Winston-Salem, North Carolina
  - Novartis Investigative Site, Fargo, North Dakota
  - Novartis Investigative Site, Cincinnati, Ohio
  - Novartis Investigative Site, Cleveland, Ohio
  - Novartis Investigative Site, Columbus, Ohio
  - Novartis Investigative Site, Marion, Ohio
  - Novartis Investigative Site, Sylvania, Ohio
  - Novartis Investigative Site, Thornville, Ohio
  - Novartis Investigative Site, Zanesville, Ohio
  - Novartis Investigative Site, Oklahoma City, Oklahoma
  - Novartis Investigative Site, Tulsa, Oklahoma
  - Novartis Investigative Site, Eugene, Oregon
  - Novartis Investigative Site, Medford, Oregon
  - Novartis Investigative Site, Erie, Pennsylvania
  - Novartis Investigative Site, Pittsburgh, Pennsylvania
  - Novartis Investigative site, Cranston, Rhode Island
  - Novartis Investigative Site, Cumberland, Rhode Island
  - Novartis Investigative Site, Greenville, South Carolina
  - Novartis Investigative Site, Johnson City, Tennessee
  - Novartis Investigative Site, Corsicana, Texas
  - Novartis Investigative Site, Dallas, Texas
  - Novartis Investigative site, El Paso, Texas
  - Novartis Investigative Site, Fort Worth, Texas
  - Novartis Investigative Site, San Antonio, Texas
  - Novartis Investigative Site, Abingdon, Virginia
  - Novartis Investigative site, Lynchburg, Virginia
  - Novartis Investigative Site, Richmond, Virginia
  - Novartis Investigative Site, Bellingham, Washington
  - Novartis Investigative site, Spokane, Washington
  - Novartis Investigative Site, Milwaukee, Wisconsin
- Argentina (2):
  - Novartis Investigative site, Buenos Aires
  - Novartis Investigative site, Rosario
- Canada (17):
  - Novartis Investigative site, Ajax
  - Novartis Investigative site, Calgary
  - Novartis Investigative site, Gatineau
  - Novartis Investigative site, Moncton
  - Novartis Investigative site, Montreal
  - Novartis Investigative site, Niagara Falls
  - Novartis Investigative site, Ottawa
  - Novartis Investigative site, Québec
  - Novartis Investigative site, Saint Romuald
  - Novartis Investigative site, Saskatoon
  - Novartis Investigative site, Sherbrooke
  - Novartis Investigative site, St. John's
  - Novartis Investigative site, Toronto
  - Novartis Investigative site, Trois-Rivières
  - Novartis Investigative site, Vancouver
  - Novartis Investigative site, Windsor
  - Novartis Investigative site, Winnipeg
- Germany (18):
  - Novartis Investigative site, Augsburg
  - Novartis Investigative site, Bad Segeberg
  - Novartis Investigative site, Berlin
  - Novartis Investigative site, Bielefeld
  - Novartis Investigative site, Bonn
  - Novartis Investigative site, Dachau
  - Novartis Investigative site, Hamburg
  - Novartis Investigative site, Hoyerswerda
  - Novartis Investigative site, Kaufbeuren
  - Novartis Investigative site, Landsberg
  - Novartis Investigative site, Leipzig
  - Novartis Investigative site, Mainz
  - Novartis Investigative site, München
  - Novartis Investigative site, Oranienburg
  - Novartis Investigative site, Oschersleben
  - Novartis Investigative site, Potsdam
  - Novartis Investigative site, Ratingen
  - Novartis Investigative site, Steinfurt-Borghorst
- India (12):
  - Novartis Investigator Site, Bangalore
  - Novartis Investigative Site, Chennai
  - Novartis Investigative Site, Coimbatore
  - Novartis Investigator Site, Coimbatore
  - Novartis Investigator Site, Hyderabaad
  - Novartis Investigator Site, Indore
  - Novartis Investigator Site, Jaipur
  - Novartis Investigator Site, Kolkata
  - Novartis Investigator Site, Ludhiana
  - Novartis Investigative Site, Mumbai
  - Novartis Investigator Site, Panjim
  - Novartis Investigator Site, Trivandrum
- Italy (14):
  - Novartis Investigator Site, Bologna
  - Novartis Investigator Site, Busto Arsizio
  - Novartis Investigator Site, Catania
  - Novartis Investigator Site, Catanzaro
  - Novartis Investigator Site, Crema
  - Novartis Investigator Site, Ferrara
  - Novartis Investigator Site, Florence
  - Novartis Investigator Site, Messina
  - Novartis Investigator Site, Milan
  - Novartis Investigator Site, Pisa
  - Novartis Investigator Site, Roma
  - Novartis Investigator Site, Rozzano
  - Novartis Investigator Site, Siena
  - Novartis Investigator Site, Sottomarina
- Spain (25):
  - Novartis Investigator Site, A Coruña
  - Novartis Investigator Site, Alicante
  - Novartis Investigator Site, Alzira
  - Novartis Investigator Site, Barcelona
  - Novartis Investigator Site, Burgos
  - Novartis Investigator Site, Córdoba
  - Novartis Investigator Site, Girona
  - Novartis Investigator Site, Gladakano
  - Novartis Investigator Site, Jerez de Frontera
  - Novartis Investigator Site, Las Palmas de Gran Canaria
  - Novartis Investigator Site, Las Palmas de Gran Canarias
  - Novartis Investigator Site, Lugo
  - Novartis Investigator Site, Madrid
  - Novartis Investigator Site, Málaga
  - Novartis Investigator Site, Ourense
  - Novartis Investigator Site, Oviedo
  - Novartis Investigator Site, Palma de Mallorca
  - Novartis Investigator Site, Ponferrada
  - Novartis Investigative Site, Pontevedra
  - Novartis Investigator Site, Port de Sagunt
  - Novartis Investigative Site, Seville
  - Novartis Investigator Site, Valencia
  - Novartis Investigator Site, Vic
  - Novartis Investigator Site, Vila-real
  - Novartis Investigative Site, Zaragoza
- Sweden (6):
  - Novartis Investigative Site, Gothenburg
  - Novartis Investigator Site, Jönköping
  - Novartis Investigative Site, Lidingö
  - Novartis Investigative Site, Luleå
  - Novartis Investigator Site, Luleå
  - Novartis Investigator Site, Lund
- Turkey (Türkiye) (3):
  - Novartis Investigative Site, Kartal/Istanbul
  - Novartis Investigator Site, Mersin
  - Novartis Investigator Site, Yenisehir/Izmir

REFERENCES:
- [Derived] Chapman KR, Rennard SI, Dogra A, Owen R, Lassen C, Kramer B; INDORSE Study Investigators. Long-term safety and efficacy of indacaterol, a long-acting beta(2)-agonist, in subjects with COPD: a randomized, placebo-controlled study. Chest. 2011 Jul;140(1):68-75. doi: 10.1378/chest.10-1830. Epub 2011 Feb 24. PMID 21349928

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is an extension study to core study stage 2: CQAB149B2335S (NCT00463567).
Groups:
- Indacaterol 300 µg: Indacaterol 300 µg once-daily (o.d.) via SDDPI. The short acting (beta) β2-agonist (SABA) salbutamol/albuterol was available for rescue use throughout the study.
Period: Overall Study
Arm/Group | Indacaterol 150 µg | Indacaterol 300 µg | Placebo
Started | 144 | 146 | 125
Safety/ITT: Received Study Drug | 144 | 146 | 124 (One patient did not take study medication.)
Completed | 126 | 135 | 105
Not Completed | 18 | 11 | 20
Not completed — Adverse Event | 4 | 1 | 6
Not completed — Lack of Efficacy | 0 | 0 | 2
Not completed — Participant no longer needs study drug | 0 | 0 | 1
Not completed — Withdrawal by Subject | 10 | 3 | 6
Not completed — Lost to Follow-up | 2 | 2 | 2
Not completed — Administrative problems | 1 | 1 | 2
Not completed — Death | 0 | 1 | 1
Not completed — Protocol Deviation | 1 | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Indacaterol 150 µg | Indacaterol 300 µg | Placebo | Total
Number analyzed (Participants) | 144 | 146 | 124 | 414
Age Continuous [Mean (Standard Deviation); unit: years] — All Baseline Measures were based on the safety population consisting of all participants who received at least one dose of study drug in the extension study.
  years | 62.5 (9.52) | 62.5 (9.00) | 62.8 (9.18) | 62.6 (9.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 60 | 43 | 160
  Male | 87 | 86 | 81 | 254

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants With a Clinically Notable Pulse Rate During 52 Weeks of Treatment With Indacaterol 150 µg or 300 µg Compared to Placebo
Description: The number of participants with newly occurring or worsening clinically notable vital sign: Pulse Rate in beats per minute (bpm) at anytime post baseline (BL) by treatment.
  Low Pulse Rate was defined as a pulse rate: <40 bpm or <= to 50 bpm and a decrease from baseline >= to 15 bpm.
  High Pulse Rate was defined as a pulse rate: >130 bpm or >= to 120 bpm and an increase from baseline >= to 15 bpm.
Time Frame: Up to 52 weeks
Population: Extension safety population consisting of all participants who received at least one dose of study drug in the extension study.
Measure: Number; unit: Participants
Arm/Group | Indacaterol 150 µg | Indacaterol 300 µg | Placebo
Number analyzed (Participants) | 144 | 146 | 124
Participants
  Low Pulse Rate | 3 | 3 | 2
  High Pulse Rate | 0 | 1 | 0

2. Secondary Outcome: Trough Forced Expiratory Volume in 1 Second (FEV1) at Week 52 of Treatment
Description: Spirometry was conducted according to internationally accepted standards. The trough FEV1 was defined as the average of the FEV1 measurements taken at 23 hours 10 minutes and 23 hours 45 minutes post dose at week 52. The mixed model used baseline FEV1 as well as FEV1 reversibility components as covariates.
Time Frame: Week 52
Population: Participants from the Extension Intent-to-treat population (consisting of all participants who received at least one dose of study drug) for whom data was available for this Outcome Measure. Missing data was imputed Last Observation Carried Forward.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Indacaterol 150 µg | Indacaterol 300 µg | Placebo
Number analyzed (Participants) | 125 | 133 | 104
Liters | 1.44 (0.034) | 1.45 (0.032) | 1.27 (0.037)

3. Primary Outcome: The Number of Participants With a Clinically Notable Systolic Blood Pressure During 52 Weeks of Treatment With Indacaterol 150 µg or 300 µg Compared to Placebo
Description: The number of participants with newly occurring or worsening clinically notable vital sign: Systolic Blood Pressure (mmHg) at anytime post baseline (BL) by treatment.
  A Low Systolic Blood Pressure was defined as a systolic blood pressure measurement: <75 mmHg or <= to 90 mmHg and a decrease from baseline >= to 20 mmHg.
  A High Systolic Blood Pressure was defined as a systolic blood pressure measurement: >200 mmHg or >= to 180 mmHg and an increase from baseline >= to 20 mmHg.
Time Frame: Up to 52 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Indacaterol 150 µg | Indacaterol 300 µg | Placebo
Number analyzed (Participants) | 144 | 146 | 124
participants
  Low Systolic Blood Pressure | 2 | 2 | 2
  High Systolic Blood Pressure | 1 | 2 | 2

4. Primary Outcome: The Number of Participants With a Clinically Notable Diastolic Blood Pressure During 52 Weeks of Treatment With Indacaterol 150 µg or 300 µg Compared to Placebo
Description: The number of participants with newly occurring or worsening clinically notable vital sign: Diastolic Blood Pressure (mmHg) at anytime post baseline (BL) by treatment.
  A Low Diastolic Blood Pressure was defined as a diastolic blood pressure measurement: <40 mmHg or <= to 50 mmHg and a decrease from baseline >= to 15 mmHg.
  A High Diastolic Blood Pressure was defined as a diastolic blood pressure measurement: >115 mmHg or >= to 105 mmHg and an increase from baseline >= to 15 mmHg.
Time Frame: Up to 52 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Indacaterol 150 µg | Indacaterol 300 µg | Placebo
Number analyzed (Participants) | 144 | 146 | 124
participants
  Low Diastolic Blood Pressure | 6 | 3 | 2
  High Diastolic Blood Pressure | 1 | 0 | 2

5. Primary Outcome: The Number of Participants With a Clinically Notable QTc Interval Value During 52 Weeks of Treatment With Indacaterol 150 µg or 300 µg Compared to Placebo
Description: The number of participants with newly occurring or worsening clinically notable QTc Interval value at anytime post baseline.
  The QTc interval is calculated using Fridericia's formula: QTc= QT/cube root RR. QTc is the interval between the Q and T waves corrected for heart rate and RR is the interval between two R waves in milliseconds (ms).
  Notable QTC interval= >450 ms for males and >470 ms for females. The maximum QTC increase from pre to post dose at any time during the study was also tabulated with absolute and relative frequencies for categories 30- 60 ms and >60 ms.
Time Frame: Up to 52 weeks
Population: as for outcome 1
Measure: Number; unit: participant
Arm/Group | Indacaterol 150 µg | Indacaterol 300 µg | Placebo
Number analyzed (Participants) | 144 | 146 | 124
participant
  Notable QTc | 10 | 9 | 11
  QTc increase from BL: 30-60 ms | 28 | 30 | 30
  QTc increase from BL: >60 ms | 1 | 1 | 1

6. Primary Outcome: Serum Potassium (mmol/L) 1 Hour Post-dose at Weeks 12, 26, 36, 44 and 52
Description: The least squares mean of the serum potassium in mmol/L at weeks 12, 26, 36, 44 and 52. Mixed model used baseline serum potassium as a covariate.
Time Frame: Weeks 12, 26, 36, 44 and 52
Population: Extension safety population consisting of all participants who received at least one dose of study drug in the extension study. "n" in the categories is the number of participants with data at the given time point for each treatment.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Indacaterol 150 µg | Indacaterol 300 µg | Placebo
Number analyzed (Participants) | 144 | 146 | 124
mmol/L
  Week 12 (n=140, 138, 115) | 4.45 (0.045) | 4.50 (0.044) | 4.45 (0.050)
  Week 26 (n=135, 141, 114) | 4.53 (0.049) | 4.53 (0.047) | 4.55 (0.053)
  Week 36 (n=132, 133, 109) | 4.46 (0.051) | 4.49 (0.050) | 4.55 (0.057)
  Week 44 (n=129, 130, 103) | 4.52 (0.050) | 4.51 (0.048) | 4.55 (0.055)
  Week 52 (n=121, 129, 97) | 4.42 (0.053) | 4.54 (0.050) | 4.49 (0.059)

7. Primary Outcome: Blood Glucose (mmol/L) 1 Hour Post Dose at Weeks 12, 26, 36, 44 and 52
Description: The least squares mean of the blood glucose in mmol/L at weeks 12, 26, 36, 44 and 52. Mixed model used baseline blood glucose as a covariate.
Time Frame: Weeks 12, 26, 36, 44 and 52
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Indacaterol 150 µg | Indacaterol 300 µg | Placebo
Number analyzed (Participants) | 144 | 146 | 124
mmol/L
  Week 12 (n=142, 140, 118) | 5.50 (0.139) | 5.59 (0.134) | 5.18 (0.150)
  Week 26 (n=137, 143, 118) | 5.93 (0.169) | 5.77 (0.160) | 5.49 (0.180)
  Week 36 (n=134, 136, 111) | 5.81 (0.156) | 5.75 (0.151) | 5.66 (0.171)
  Week 44 (n=131, 133, 105) | 5.70 (0.189) | 5.88 (0.176) | 5.60 (0.205)
  Week 52 (n=123, 131, 99) | 5.93 (0.201) | 5.70 (0.189) | 5.55 (0.221)

8. Secondary Outcome: Quality of Life Assessment With St George's Respiratory Questionnaire (SGRQ) Total Score at Weeks 36, 44 and 52
Description: The least squares mean of the SGRQ total score at weeks 36, 44 and 52. Mixed model used for analysis used baseline SGRQ total score as well as FEV1 reversibility components as covariates.
  SGRQ is a health related quality of life questionnaire consisting of 50 items in three domains: symptoms, activity and impacts. The total score is 0 to 100 with a higher score indicating poorer health. A difference from placebo of -4 in the least squares mean SGRQ total score is considered clinically relevant.
Time Frame: Weeks 36, 44 and 52
Population: Extension Intent-to-treat population consisting of all participants who received at least one dose of study drug. "n" in each of the categories is the number of participants with data at the given time point. Missing data were imputed using LOCF but not by more than 14 weeks and not by carrying forward scores within 4 weeks of treatment start.
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | Indacaterol 150 µg | Indacaterol 300 µg | Placebo
Number analyzed (Participants) | 144 | 146 | 124
Score on a Scale
  Week 36 (n=138, 137, 113) | 36.62 (1.767) | 36.37 (1.695) | 39.56 (1.913)
  Week 44 (n= 128, 133, 109) | 35.98 (1.883) | 36.18 (1.739) | 41.67 (2.001)
  Week 52 (n=126, 132, 104) | 35.97 (1.826) | 37.49 (1.721) | 39.19 (2.004)

ADVERSE EVENTS:
Time Frame: 26 weeks
Description: Safety population consisting of all participants who received at least one dose of study drug in the extension study.
Arm/Group | Indacaterol 150 µg | Indacaterol 300 µg | Placebo
Serious Adverse Events (participants affected / at risk) | 15/144 | 18/146 | 13/124
Other Adverse Events (participants affected / at risk) | 86/144 | 91/146 | 67/124
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Indacaterol 150 µg (N=144) | Indacaterol 300 µg (N=146) | Placebo (N=124)
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0
Cardiovascular disorder (Cardiac disorders) | 0 | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1 | 1
Sick sinus syndrome (Cardiac disorders) | 0 | 1 | 0
Endocardial fibroelastosis (Congenital, familial and genetic disorders) | 0 | 0 | 1
Cataract (Eye disorders) | 0 | 1 | 0
Faecaloma (Gastrointestinal disorders) | 0 | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0
Appendicitis perforated (Infections and infestations) | 1 | 0 | 0
Infection (Infections and infestations) | 1 | 0 | 0
Lobar pneumonia (Infections and infestations) | 0 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 1
Pelvic abscess (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0 | 2
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Cerebellar infarction (Nervous system disorders) | 0 | 0 | 1
Syncope (Nervous system disorders) | 1 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 4 | 5 | 3
Laryngeal leukoplakia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary calcification (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Intermittent claudication (Vascular disorders) | 0 | 1 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 0 | 0
Peripheral vascular disorder (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Indacaterol 150 µg (N=144) | Indacaterol 300 µg (N=146) | Placebo (N=124)
Diarrhoea (Gastrointestinal disorders) | 5 | 5 | 7
Nausea (Gastrointestinal disorders) | 4 | 6 | 7
Bronchitis (Infections and infestations) | 5 | 9 | 9
Influenza (Infections and infestations) | 8 | 5 | 3
Lower respiratory tract infection (Infections and infestations) | 5 | 11 | 8
Nasopharyngitis (Infections and infestations) | 24 | 26 | 19
Sinusitis (Infections and infestations) | 9 | 11 | 3
Upper respiratory tract infection (Infections and infestations) | 17 | 20 | 10
Urinary tract infection (Infections and infestations) | 5 | 8 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 8 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 4 | 7
Muscle spasms (Musculoskeletal and connective tissue disorders) | 12 | 4 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 5 | 8 | 1
Headache (Nervous system disorders) | 15 | 7 | 5
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 34 | 36 | 33
Cough (Respiratory, thoracic and mediastinal disorders) | 17 | 15 | 8
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 | 4 | 6
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 10 | 10 | 2
Hypertension (Vascular disorders) | 6 | 3 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.